CLINICAL TRIAL: NCT01514695
Title: Fentanyl Use for Sedation in Esophagogastroduodenoscopy (FUSE): a Phase 4, Randomized, Double-blind, Placebo-controlled Trial of Fentanyl Added to Midazolam Compared to Midazolam Alone for Sedation in Routine Upper Endoscopy
Brief Title: Fentanyl Use for Sedation in Esophagogastroduodenoscopy
Acronym: FUSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Khurram Khan, Assistant Professor of Medicine, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R.P. 11-3611
Record Dates: First submitted 2012-01-11; First posted 2012-01-23 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Endoscopy
Keywords: endoscopy; sedation; opioid; narcotic
MeSH Terms: interventions — Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl (Experimental): Fentanyl arm
  Interventions: Drug: Midazolam; Drug: Fentanyl
- Placebo (Placebo Comparator): Placebo of identical appearance
  Interventions: Drug: Midazolam; Other: Placebo

INTERVENTIONS:
Drug: Midazolam — Starting with 1mg intravenously in all patients. More can be added at the discretion of the physician as needed for sedation.
Drug: Fentanyl — 100mcg intravenously given in 2mL syringe at start of procedure
  Arms: Fentanyl
Other: Placebo — One dose of saline (2ml)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether conscious sedation with a narcotic and sedative (in combination) is as efficacious as a sedative alone for elective upper endoscopy to achieve optimal patient comfort and ease of procedure.

DETAILED DESCRIPTION:
Upper endoscopy is a valuable procedure that involves a camera advanced from the mouth into the intestines. It is a routine test and considered very safe. However, patients can experience discomfort from air insufflation in the stomach and unpleasantness due to gagging during the procedure. Conscious sedation with medications like sedatives and narcotics are used to improve patient satisfaction and enhance physician ability to perform an optimal examination. The choice of drugs used for sedation in upper endoscopy varies by endoscopist and the goal is always to use the lowest dose possible to achieve the best examination. Combination therapy (with a sedative & narcotic) may increase the adverse effect profile compared to a sedative alone and not improve the overall experience of the physician or patient. The goal of our study is to assess in randomized, double-blind, placebo controlled study, the effect of using a narcotic (fentanyl) and sedative (midazolam) for sedation compared to a sedative (midazolam) alone.

ELIGIBILITY:
Inclusion Criteria:

* outpatient elective upper endoscopy
* age 18-65
* able to give consent

Exclusion Criteria:

* mental incompetency
* pregnancy
* weight <55kg or 110 lbs
* emergent procedures,
* known hypersensitivity or allergy to fentanyl or midazolam
* chronic use of benzodiazepines or opioids
* patients known a priori to require therapeutic interventions in conjunction with their EGD
* patients to have major cardiorespiratory comorbidities, obstructive sleep apnea, liver cirrhosis, or renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with the level of sedation and comfort during the procedure on an analog scale | Within 72 hours of procedure
  Level of satisfaction is obtained by telephone the following day, and up to 72 hours after the procedure.

SECONDARY OUTCOMES:
Physician satisfaction with the level of sedation and ease of procedure based on a visual analog scale | Following procedure up to time of discharge (average of 45 minutes after procedure started)
Patient willingness to repeat procedure | Asked within 72 hours of procedure
Presence of significant retching | Following procedure up to time of discharge (average of 45 minutes after procedure started)
  Recorded by physician completing procedure
Presence of adverse events | Following procedure up to time of discharge (average of 45 minutes after procedure started)
  Any adverse event during procedure up until patient leaves endoscopy unit

CONTACTS AND LOCATIONS:
Overall Officials: Khurram J Khan, MD, BSc, MSc, Principal Investigator — St Joseph's Healthcare Hamilton, McMaster University
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada